CLINICAL TRIAL: NCT04456010
Title: Assessing the Perception and the Personal Experience of the COVID19 Pandemic Among Infertile Couples Undergoing Assisted Reproductive Treatment (ART)
Brief Title: COVID-19 in ART: Perception and Experience
Acronym: COVAPEX
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0351
Record Dates: First submitted 2020-06-15; First posted 2020-07-02 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID19; Fertility Issues; ART
Keywords: fertility; risk perception; emotional experience
MeSH Terms: conditions — COVID-19; Infertility | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile couple: Infertile couple who had a fertility treatment prescribed during the past 9 months which was not completed yet.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Eligible patients will be selected from our electronical database and invited via email to participate.

SUMMARY:
Non-urgent medical care, such as fertility treatments, has been massively postponed during the past weeks due to the COVID19 pandemic. The lockdown and the closure of IVF centers might cause anxiety and depression among infertile couples, who are already exposed to the distressing experience of infertility and for whom the wait for a baby already appears unending. Few data are available regarding the impact of SARS-CoV-2 on pregnant women and foetus, or on fertility.

This study aims to assess the views of infertile couple regarding the potential risks of COVID during their fertility treatment and their personal experience of the COVID pandemic and their expectation for further treatment .

ELIGIBILITY:
Inclusion criteria:

- Men and women who had a fertility treatment prescribed during the past 9 months in our Fertility department

Exclusion criteria:

* Patient attending for a fertility preservation
* Patient attending for a preimplantation genetic testing (PGT-M or PGT-SR)
* Patient not fluent in French

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile couple (male and female) who had a fertility treatment prescribed during the past 9 months (prescription after October 1st, 2019) in the fertility department of Montpellier Hospital
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Personal experience of the COVID19 pandemic and the discontinuation of their fertility treatment pandemic and the discontinuation | 1 day
  Personal experience of the COVID19 pandemic and the discontinuation of their fertility treatment, via a survey

SECONDARY OUTCOMES:
Risk assessment | 1 day
  . Risk assessment by the patient, via a survey, regarding SARS-CoV-2 during a fertility treatment or during pregnancy. Perception of the risks linked to SARS-CoV-2 during their fertility treatment or during a pregnancy
Patients'expectations regarding the management of an abrupt closure of the fertility center | 1 day
  Patients'expectations regarding the management of an abrupt closure of the fertility center, via a survey

CONTACTS AND LOCATIONS:
Overall Officials: Noémie Ranisavljevic, M.D., Ph.D, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC